CLINICAL TRIAL: NCT03496610
Title: Intraoperative Surgical Wound Infiltration vs Quadratus Lumborum (QL) Block for Post-operative Pain Control After Nephrectomy in Living Donor Kidney Transplant Patients
Brief Title: Surgeon Infiltration QL Block Comparison
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00087144
Record Dates: First submitted 2018-04-05; First posted 2018-04-12 (Actual); Results first posted 2024-03-05 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-02

CONDITIONS: Quadratus Lumborum Block; Surgical Wound Infiltration
Keywords: Bupivacaine; Living donor nephrectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Quadratus Lumborum (QL) Block (Active Comparator): Patients will receive a bilateral ultrasound guided QL block by the anesthesia team.
  Interventions: Procedure: QL Block
- Surgical wound infiltration (Active Comparator): Patients will receive 266 mg of liposomal bupivacaine mixed with 50 mg non-liposomal bupivacaine infiltrated into the wound by the surgeon.
  Interventions: Drug: Liposomal Bupivicaine

INTERVENTIONS:
Drug: Liposomal Bupivicaine — Patient will receive liposomal bupivicaine mixed with non-liposomal bupivicaine directly to wound
  Arms: Surgical wound infiltration
Procedure: QL Block — Patient will receive ultrasound guided QL Block
  Arms: Quadratus Lumborum (QL) Block

SUMMARY:
The purpose of this study is to learn if using a Quadratus Lumborum (QL) plane injection technique (also called a "nerve block") that numbs the nerves going to the abdominal area improve pain control after surgery compared to administration of local anesthetic directly to the surgical incision. The QL block technique uses a numbing solution (local anesthetics) that is injected next to nerves located along muscles in the back to reduce pain. This block will not affect movement in the leg and/or make the legs weak. Some institutions, including Duke, use the QL block for patients having various abdominal surgeries, with the hope of providing good pain relief combined with improved mobility after surgery.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* ASA 1-2 patients undergoing living donor nephrectomy

Exclusion Criteria:

* ASA 3 or 5
* Diagnosis of chronic pain
* Daily chronic opioid use (over 3 months of continuous opioid use)
* Inability to communicate pain scores or need for analgesia
* Infection at the site of block placement
* Pregnant women (as determined by standard of care day-of surgery urine bHCG)
* Intolerance/allergy to local anesthetics
* Weight <50 kg
* Suspected or known addiction to or abuse of illicit drug(s), prescription medicine(s), or alcohol within the past 2 years
* Uncontrolled anxiety, schizophrenia, or other psychiatric disorder that, in the opinion of the investigator, may interfere with study assessments or compliance
* Current or historical evidence of any clinically significant disease or condition that, in the opinion of the investigator, may increase the risk of surgery or complicate the subject's postoperative course

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2021-01-25 (Actual); Primary Completion 2023-02-23 (Actual); Study Completion 2023-02-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hector Martinez-Wilson, MD, Principal Investigator — Duke University
Locations (1):
- Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Quadratus Lumborum (QL) Block | Surgical Wound Infiltration
Started | 24 | 20
Completed | 19 | 18
Not Completed | 5 | 2
Not completed — Lost to Follow-up | 3 | 2
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: The number of participants in the QL group excludes two subjects-- one subject who voluntarily withdrew and one who was withdrawn by the PI for a surgical site infection.
Groups:
- Total: Total of all reporting groups
Arm/Group | Quadratus Lumborum (QL) Block | Surgical Wound Infiltration | Total
Number analyzed (Participants) | 22 | 20 | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.59 (14.41) | 47.90 (12.51) | 45.25 (13.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 13 | 28
  Male | 7 | 7 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 22 | 19 | 41
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 4 | 10
  White | 16 | 16 | 32
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 22 | 20 | 42

OUTCOME MEASURES:

1. Primary Outcome: Opioid Consumption in Oral Morphine Milliequivalents for the First 24 Hours After Surgery (Defined as 24 Hours After the Anesthesia End Time)
Time Frame: 24 hours postoperatively
Population: This analysis excludes two subjects who were originally enrolled in the QL group--one subject who voluntarily withdrew and one who was withdrawn by the PI for a surgical site infection.
Measure: Median (Inter-Quartile Range); unit: oral morphine equivalents in milligrams
Arm/Group | Quadratus Lumborum (QL) Block | Surgical Wound Infiltration
Number analyzed (Participants) | 22 | 20
oral morphine equivalents in milligrams | 17.50 [6.88 to 33.88] | 21.25 [7.50 to 46.88]
Statistical Analysis 1: Comparison: Quadratus Lumborum (QL) Block vs Surgical Wound Infiltration; Wilcoxon Rank Sum test performed given non-normal distribution of data by Shapiro Wilks Test. Null hypothesis is that there is no difference in oral morphine equivalent consumption between the two groups in the first 24hrs after surgery. Original sample size calculation based on α=0.05, β=0.8, difference in means=2, and effect size of 1.0; Test type: Superiority; p = 0.81, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Self-reported Numeric Pain Scores on Postoperative Day Seven
Description: Pain was measured on a self-reported scale of 0-10, where 0=no pain and 10=worst imaginable pain. Scores were gathered by phone on postoperative day 7.
Time Frame: Postoperative day 7
Population: This analysis excludes two subjects who were originally enrolled in the QL group--one subject who voluntarily withdrew and one who was withdrawn by the PI for a surgical site infection. Five subjects (3 in the QL group and 2 in the infiltration group) were not reachable by phone on postoperative day 7 and were therefore excluded from this analysis.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Quadratus Lumborum (QL) Block | Surgical Wound Infiltration
Number analyzed (Participants) | 19 | 18
score on a scale | 2 [1 to 3] | 1 [1 to 2]
Statistical Analysis 1: Comparison: Quadratus Lumborum (QL) Block vs Surgical Wound Infiltration; Wilcoxon Rank Sum test performed with α=0.05. The null hypothesis is that there is no difference between the two groups in pain on postoperative day 7; Test type: Superiority; p = 0.40, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Worst Bloating Severity in the First Postoperative Week
Description: Bloating severity scores were gathered daily by phone interview for the first week postoperatively. Bloating severity was assessed on a scale of 1-5, where 1= not at all severe and 5=very much. The highest severity score reported during the week was collected for this outcome measure.
Time Frame: First seven days postoperatively
Population: This analysis excludes two subjects who were originally enrolled in the QL group--one subject who voluntarily withdrew and one who was withdrawn by the PI for a surgical site infection. Five subjects (3 in the QL group and 2 in the infiltration group) were not reachable by phone and were therefore excluded from this analysis.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Quadratus Lumborum (QL) Block | Surgical Wound Infiltration
Number analyzed (Participants) | 19 | 18
score on a scale | 4 [3 to 5] | 4 [2.75 to 5]
Statistical Analysis 1: Comparison: Quadratus Lumborum (QL) Block vs Surgical Wound Infiltration; Wilcoxon Rank Sum test performed with α=0.05. The null hypothesis is that there is no difference in bloating severity between the two groups; Test type: Superiority; p = 0.74, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Self-reported Ability to Walk for 15 Minutes Without Any Difficulty Within the First Postoperative Week
Description: Physical function was assessed by daily phone interview during the first postoperative week. Subjects were asked to assess their ability to go for a walk of at least 15 minute on a scale of 1-5 with 1=unable to do and 5= able to do without any difficulty. For this outcome, the number of subjects who reported being able to go for a walk of at least 15 minutes "without any difficulty" at any time during the first postoperative week is reported.
Time Frame: First seven days postoperatively
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Quadratus Lumborum (QL) Block | Surgical Wound Infiltration
Number analyzed (Participants) | 19 | 18
Participants | 10 | 12
Statistical Analysis 1: Comparison: Quadratus Lumborum (QL) Block vs Surgical Wound Infiltration; Compared using the Likelihood ratio test with α=0.05. The null hypothesis was that there is no difference between the groups; Test type: Other; p = 0.38, Chi-squared; Degrees of freedom = 1

ADVERSE EVENTS:
Time Frame: Up to 7 days
Arm/Group | Quadratus Lumborum (QL) Block | Surgical Wound Infiltration
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/20
Other Adverse Events (participants affected / at risk) | 0/24 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-11-09): https://cdn.clinicaltrials.gov/large-docs/10/NCT03496610/Prot_SAP_000.pdf